CLINICAL TRIAL: NCT01472354
Title: Feasibility of a HCV Decision-Making Intervention Among HIV-infected Adults
Brief Title: Feasibility of a Hepatitis C Virus (HCV) Decision-Making Intervention Among HIV-infected Adults
Acronym: LEAP-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Carol Bova, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S61110000013230; R21NR011132 (NIH)
Record Dates: First submitted 2011-08-02; First posted 2011-11-16 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Hepatitis c
Keywords: HIV; Hepatitis C; Decision-Making; chronic
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care referral to specialist (No Intervention): Subjects are referred for education, counseling and evaluation for HCV treatment to a specialty health care provider
- LEAP-C Group Intervention (Experimental): 4-week group intervention to help HIV/HCV co-infected patients reframe negative appraisals associated with HCV treatment to decrease decisional conflict, increase HCV knowledge, improve communication
  Interventions: Behavioral: Leap-c group intervention

INTERVENTIONS:
Behavioral: Leap-c group intervention — 4-week group intervention to help HIV/HCV co-infected patients reframe negative appraisals associated with hCV treatment, increase HCV knowledge, increase skills related to working with health care providers
  Other Names: LEAP-C
  Arms: LEAP-C Group Intervention

SUMMARY:
The purpose of the LEAP-C (learning, experiencing and preparing for hepatitis C treatment) study is to see if a brief (4-week) small group intervention will help people with HIV/HCV co-infection make an informed decision about Hepatitis C treatment.

DETAILED DESCRIPTION:
Chronic Hepatitis C Virus (HCV) infection is a major problem for Human Immunodeficiency Virus (HIV)-infected patients. Without HCV treatment, increasing numbers of HIV positive patients will die either from end stage liver disease or from HIV-related complications because of the inability to use antiretroviral agents due their hepatotoxicity. Major advances in understanding HCV treatment in this population have occurred within the past several years. Yet, only a small proportion of co-infected patients receive HCV treatment (approximately 15%). Moreover, few studies have explored patient decision-making related to HCV treatment in HIV co-infected patients. The major gap in our knowledge is how best to support patients as they engage in the HCV treatment decision making process with their health care provider. Therefore, the purpose of this phase II study is to test the feasibility of conducting a theoretically-derived group intervention with HIV/HCV co-infected adults to support active engagement in HCV treatment decision-making. The primary aims are to: (1) determine the feasibility of recruiting and retaining a sample of HIV/HCV co-infected adults to complete a protocol that involves randomization into the 4-week HCV Positive Life Skills group intervention or usual care and completion of two data collection interviews (at baseline and week 12), (2) establish the preliminary effect size of the HCV Positive Life Skills group intervention on HCV knowledge, decisional conflict, patient-provider communication, health-related quality of life, symptom experience and engagement with health care providers, (3) explore the capacity of the group intervention to influence HCV knowledge, decisional conflict, patient-provider communication, engagement with health care providers, health related quality of life and symptom experience and (4) describe the components of the intervention and usual care (through qualitative interviews) that are most useful for helping HIV/HCV co-infected patients engage in decision-making about HCV treatment. A mixed method approach will be used. 50 HIV/HCV co-infected participants will be randomized equally to receive either the group intervention or usual care. Then qualitative interviews, using qualitative descriptive methods, will be conducted with 10-12 participants to identify the most salient parts of the intervention and usual care that support effective decision-making about HCV treatment. The investigators will also compare the time spent with both groups, identify variability in the control condition, describe the number of subjects who start HCV treatment and further refine the intervention manual and intervention fidelity procedures in preparation for a full scale multi-site randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Men and Women (18 years of age or older) who have both HIV and chronic Hepatitis C (they need to have a detectable Hepatitis C viral load)

HIV/HCV co-infected adults who have NEVER started treatment

HIV/HCV co-infected adults who DO NOT have a MEDICAL reason that would make it dangerous to treat their hepatitis C (for example, severe cirrhosis already)

HIV/HCV co-infected adults who would be willing to be RANDOMIZED into a group session or standard of care (one on one care with a HCV provider)

Exclusion Criteria:

Non-English Speaking

Children under age 18

HCV mono-infected adults

HIV/HCV co-infected adults who have received any HCV treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Decrease in decisional conflict related to HCV treatment 12 weeks post treatment | Up to 12 weeks
  Collect data on the study sample at baseline and week 12 to determine whether the intervention decreased decisional conflict.

SECONDARY OUTCOMES:
Proportion of subjects electing HCV treatment 6 months after enrollment in the feasibility study. | 6 months
  Collect data on the study sample to determine the proportion of subjects who began HCV treatment 6 months after enrollment in the study.
Increase in knowledge related to HCV treatment 12 weeks post treatment | Up to 12 weeks
  Collect data at baseline and week 12 to determine whether the intervention improved HCV-related knowledge.
Increase in communication between subject and health care provider from baseline to week 12. | Up to 12 weeks
  Collect data on the study sample at baseline and week 12 to determine whether the intervention has improved the subjects' perception of communication with their health care provider.
Increase in subjects' health related quality of life from baseline to 12 weeks after study enrollment | Up to 12 weeks
  Collect data on the study sample at baseline and week 12 to determine whether the intervention has improved subjects' perception of health related quality of life.
Number of symptoms experienced by HCV infected subjects from baseline to week 12 | Up to 12 weeks
  Collect data on the study sample at baseline and week 12 to determine whether the intervention has decreased the number of symptoms experienced by the research subjects.
Severity of symptoms experienced by HCV infected subjects from baseline to week 12 | Up to 12 weeks
  Collect data on the study sample at baseline and week 12 to determine whether the intervention has decreased the severity of symptoms experienced by the research subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Graduate School of Nursing, Worcester, Massachusetts, United States